CLINICAL TRIAL: NCT00262184
Title: A Taiwan Isoflavone Multicenter Study (TIMS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taiwan Biotech Co., Ltd. (Industry); Genovate Biotechnology Co., Ltd., (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GE-PP02; NCT00154908 (obsolete NCT alias)
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2005-12-06 (Estimated); Status verified 2005-12

CONDITIONS: Low Bone Density; Osteopenia
Keywords: Post-Menopausal osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Soybean Proteins

INTERVENTIONS:
Drug: Soy Isoflavone

SUMMARY:
Consumption of soy-based foods is associated with a number of health benefits, including lower risk of cardiovascular disease, breast and prostate cancer, attenuated menopausal symptoms and prevention of bone loss with age.

In order to investigate the effect of isoflavone on bone mineral density (BMD) and in Taiwan women with postmenopausal osteopenia, a Taiwan Isoflavone Multicentric Enrollment Study (TIMS) is designed.

DETAILED DESCRIPTION:
Consumption of soy-based foods is associated with a number of health benefits, including lower risk of cardiovascular disease, breast and prostate cancer, attenuated menopausal symptoms and prevention of bone loss with age.

In order to investigate the effect of isoflavone on bone mineral density (BMD) and in Taiwan women with postmenopausal osteopenia, a Taiwan Isoflavone Multicentric Enrollment Study (TIMS) is designed. Included in the study will be Taiwanese, postmenopausal women aged >45 and < 65 years, menopaused for at least 12 months and less than 10 years. Three medical centers will participate and enroll 140 women in every center. Inclusion will be on the basis of a lumbar bone mineral density (BMD) lower than 1 SD compared with young age women (T score) by DXA. Women with prevalent fractures (any kind of fragility fracture, vertebral or nonvertebral fracture) are excluded as well as those presenting secondary osteoporosis or having been treated with medications that could affect bone metabolism. This study is designed as a 2-year, double-blind, placebo-controlled, two-arm, parallel group study that randomizes the women to the oral administration of 300 mg isoflavone aglycone/day or placebo. All patients receive a daily supplement of 600 mg calcium and 300U of Vit D3. The primary endpoint of the study is to evaluate the effect of isoflavone aglycone on BMD. The secondary endpoint of the study will be to evaluate the effect of Isoflavone aglycone on the metabolic indicators of osteoporosis, blood pressure, blood sugar and insulin level, insulin resistance (HOMA-IR), lipid profile, markers of arthrosclerosis (adiponectin and hsCRP), myocardial infarction rate, cardiovascular mortality, cerebrovascular accident rate, cerebrovascular mortality, all cause mortality and symptomatic relief of menopausal syndrome, BMD reading will be done concomitantly by 3 experts, e.g. one from each participating center. All blood test and urine examination will be done at one center for control of quality. The blood count, biochemistry (including: GOT, GPT, BUN, creatinine), mammography, and gynecological sonography (especially uterus) will be performed to monitor the side effects.

Power calculations have been based on the hypothesis that isoflavone-treated patients would get 2.5% benefit in BMD than placebo-treated patients in postmenopausal women. Statistical tests have been designed to have a power of 80%, with a type I error equal to 5%. This study should verify the hypothesis that isoflavone significantly increase the BMD in Asian postmenopausal osteopenic women.

ELIGIBILITY:
Inclusion Criteria:

1. The postmenopausal women who menopaused for at least 12 months and less than 10 years.
2. The postmenopausal women aged >45 and < 65 years.
3. For those being done with hysterectomy and age between 50 and 60, with FSH >40 IU/l and Estradiol < 40 pg/ml.
4. Bone mineral density (BMD) of lumbar spine L2-L4 (AP view) lower than 1 SD compared with young age women (T score<-1)
5. BMI, above 18.5kg/m2 and below 30 kg/m2
6. Willingness to comply with the protocol and signed the written Informed Consent.

Exclusion Criteria:

1. Any prevalent vertebral, hip or wrist fractures.
2. Secondary osteoporosis, osteomalacia, Paget's disease of bone, multiple myeloma, or bone metastases.
3. Hormonal replacement therapy (HRT) or SERM within the previous 3 months
4. Phytoestrogen treatment within the previous 3 months
5. Fluoride treatment within the previous 6 months
6. Bisphosphate treatment within the previous 12 months
7. Calcitonin treatment within the previous 6 months
8. Any other treatment affecting the bone mineral density within the previous 6 months
9. Chronic systemic corticosteroid treatment within the previous 6 months
10. History of Gynecological cancer or breast cancer
11. Cervical smear class III or IV, according to the Bethesda system.
12. Undiagnosed vaginal bleeding.
13. Known or suspected estrogen-dependent tumors, fibroids or endometrial polyps
14. Significant or Pathological endometrial hyperplasia
15. Active major psychiatric disorders
16. Alcoholism or drug abuse
17. Known cardiovascular, cerebrovascular or peripheral vascular disorders (e.g. thrombophlebitis, thromboembolism)
18. Uncontrolled Diabetes with HbA1C > 10%
19. Uncontrolled hypertension with blood pressure > 180/100 mmHg
20. Uncontrolled hypothyroidism
21. Any renal disease with serum creatinine > 2mg/dl
22. Abnormal liver function with S-ALT and S-AST values> 2-fold upper limits

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420
Dates: Start 2004-12; Study Completion 2007-12

PRIMARY OUTCOMES:
BMD change

SECONDARY OUTCOMES:
Lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Tong-Yuan Tai, MD & PHD, Principal Investigator — NHRI
Locations (3):
- Taiwan (3):
  - National Taiwan University Hospital, Taipei, Taipei
  - Chang-hua Christian Hospital, Chang-hua
  - National Cheng-Kung University Hospital, Tainan